CLINICAL TRIAL: NCT02089269
Title: Clinical Registry on Treatment Reality and Sequential Treatments of Patients with Resectable or Locally Advanced/metastatic Pancreatic Cancer in Real-life Practice in Germany
Brief Title: Tumor Registry Pancreatic Cancer
Acronym: AMETHYST
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: iOM-01281; Tumorregister Pankreaskarzinom (Other: iOMEDICO)
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2024-10

CONDITIONS: Pancreas Cancer
Keywords: pancreatic neoplasms; neoplasms; registry; advanced pancreatic cancer; health services research; epidemiology; Germany; palliative treatment; palliative care; localized, resectable pancreatic cancer; adjuvant treatment
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: 2,200 patients with unresectable locally advanced or metastatic pancreatic cancer, treated in palliative intention
- Cohort 2: 125 patients with localized, resectable pancreatic cancer treated in neo-adjuvant or adjuvant intention

SUMMARY:
The registry aims to collect and analyse information on the antineoplastic treatment of patients with unresectable locally advanced or metastatic pancreatic cancer, treated in palliative intention (cohort 1) and patients with localized, resectable pancreatic cancer treated in neo-adjuvant or adjuvant intention (cohort 2) in daily routine practice in Germany. The registry will follow up patients for two years. It will identify common sequences of treatments used as well as changes in the treatment of the disease. Health-related quality of life will be analysed during the course of the treatment (PanLife). Based on the available data a prognostic score will be developed.

ELIGIBILITY:
Inclusion Criteria:

* resectable or locally advanced/metastatic pancreatic cancer
* 18 years and older
* Antineoplastic treatment
* Date of consent no later than 2 weeks after start of first-line treatment

Exclusion Criteria:

* No pancreatic cancer
* Below 18 years and older
* No antineoplastic treatment
* Date of consent later than 2 weeks after start of first-line treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cancer undergoing antineoplastic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 2325 (Actual)
Dates: Start 2013-12; Primary Completion 2022-04-14 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Treatment reality in Germany | over 5 years
  description of treatments selected for patients per line of therapy over the course of the project

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Hegewisch-Becker, Prof. MD, Study Chair — Outpatient Clinic, Hamburg
Locations (1):
- iOMEDICO, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hegewisch-Becker S, Aldaoud A, Wolf T, Krammer-Steiner B, Linde H, Scheiner-Sparna R, Hamm D, Janicke M, Marschner N; TPK-Group (Tumour Registry Pancreatic Cancer). Results from the prospective German TPK clinical cohort study: Treatment algorithms and survival of 1,174 patients with locally advanced, inoperable, or metastatic pancreatic ductal adenocarcinoma. Int J Cancer. 2019 Mar 1;144(5):981-990. doi: 10.1002/ijc.31751. Epub 2018 Oct 3. PMID 30006989
- [Background] Marschner N, Hegewisch-Becker S, Reiser M, von der Heyde E, Bertram M, Hollerbach SH, Kreher S, Wolf T, Binninger A, Chiabudini M, Kaiser-Osterhues A, Janicke M; TPK-Group (Tumour Registry Pancreatic Cancer). FOLFIRINOX or gemcitabine/nab-paclitaxel in advanced pancreatic adenocarcinoma: A novel validated prognostic score to facilitate treatment decision-making in real-world. Int J Cancer. 2023 Feb 1;152(3):458-469. doi: 10.1002/ijc.34271. Epub 2022 Sep 22. PMID 36053905
- [Background] Marschner N, Haug N, Hegewisch-Becker S, Reiser M, Dorfel S, Lerchenmuller C, Linde H, Wolf T, Hof A, Kaiser-Osterhues A, Potthoff K, Janicke M; TPK-Group (Tumour Registry Pancreatic Cancer). Head-to-head comparison of treatment sequences in advanced pancreatic cancer-Real-world data from the prospective German TPK clinical cohort study. Int J Cancer. 2024 Nov 1;155(9):1629-1640. doi: 10.1002/ijc.35071. Epub 2024 Jul 2. PMID 38956837